CLINICAL TRIAL: NCT01286493
Title: Immune Response After Booster Vaccination in HIV - Infected Patients Who Ever Received Rabies Primary Vaccination
Brief Title: Immune Response After Booster Vaccination in HIV - Infected Patients Who Received Rabies Primary Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal investigator, Queen Saovabha Memorial Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC5303
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: HIV; Rabies
Keywords: HIV; booster; rabies; immune response
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rabies vaccines on day 0 and 3 (Experimental): Cell culture Rabies vaccines on day 0 and 3
  Interventions: Biological: rabies vaccines on day 0 and 3

INTERVENTIONS:
Biological: rabies vaccines on day 0 and 3 — All subjects would receive conventional intramuscular booster rabies vaccination on day 0 and 3. Their blood would be drawn for rabies neutralizing antibody on day 0,7,14,30,90,180,360

SUMMARY:
Booster rabies vaccination in HIV - infected patients who have ever received rabies primary vaccination could improve their immune response to this kind of vaccine.

DETAILED DESCRIPTION:
The investigators have learned from the previous studies that some HIV-infected patients especially those with low CD4+ T-lymphocyte count had poor antibody response to rabies vaccination. Because of the role of the memory B cell, the investigators hypothesized that primary rabies immunization in HIV-infected patients could rise rapid anamnestic antibody response to ones after booster vaccination in case of re-exposure of rabies occur despite of their immunocompromised state.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients 18-60 years of age
* Ever received primary rabies immunization

Exclusion Criteria:

* currently have any active opportunistic infections
* have received blood or blood product within previous 3 months
* history of allergy to vaccine or any vaccine components
* currently received anti-malarial drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: http://www.saovabha.com/th/academic.asp — http://www.saovabha.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Rabies Vaccines on Day 0 and 3: Cell culture Rabies vaccines on day 0 and 3
  rabies vaccines on day 0 and 3: All subjects would receive conventional intramuscular booster rabies vaccination on day 0 and 3. Their blood would be drawn for rabies neutralizing antibody on day 0,7,14,28,90,180,360
Period: Overall Study
Arm/Group | Rabies Vaccines on Day 0 and 3
Started | 33
Completed | 30
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Preliminary study
Arm/Group | Rabies Vaccines on Day 0 and 3
Number analyzed (Participants) | 33
Age, Continuous [Median (Standard Deviation); unit: years] | 43 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Region of Enrollment [Number; unit: participants]
  Thailand | 33
CD4+ T lymphocyte counts [Median (Full Range); unit: cell/mm^3] | 489 [94 to 1120]

OUTCOME MEASURES:

1. Primary Outcome: Rabies Neutralizing Antibody Titers
Description: Rabies Neutralizing Antibody titers(RNab)of HIV-infected patients who receive booster rabies vaccination would be measured by Rapid Fluorescent Focus Inhibition Test(RFFIT) method at day 0, 7, 14, 28, 90,180 and 360. RNab level above 0.5 IU/ml indicate acceptable protective antibody response.
  for 7 times in 1 year.
Time Frame: Day 360
Population: As preliminary study, the number of participants was estimated to be above 15 - 20 cases.
Measure: Geometric Mean (Full Range); unit: IU/ml
Arm/Group | Rabies Vaccines on Day 0 and 3
Number analyzed (Participants) | 33
IU/ml | 8.48 [0.50 to 218.10]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rabies Vaccines on Day 0 and 3
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

LIMITATIONS AND CAVEATS:
Small sample size heterogeneous characteristics of participants Use only CD4+ T lymphocyte counts as the only immunologic surrogate marker

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes